CLINICAL TRIAL: NCT03805646
Title: A Mobile Phone-based Triage Tool to Identify Discharged Trauma Patients in Need of Further Care in Cameroon
Brief Title: Mobile Phone-administered Triage Tool to Followup on Discharged Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Buea (Other)
Responsible Party: Principal Investigator, Catherine Juillard, MD, MPH, Associate Professor In-Residence, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GRANT12763845
Record Dates: First submitted 2019-01-11; First posted 2019-01-16 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Wounds and Injury
Keywords: Aftercare; Telemedicine; Africa South of the Sahara
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: None of the interventional study model categories aptly describe the study. The step-wedge design of the study means each site has historical controls; the only thing determining whether an individual receives the intervention or not is time (that is, whether the hospital site s/he was admitted to happens to be in the pre-intervention/baseline data collection phase or the intervention phase).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Mobile Phone-administered Triage Tool (No Intervention): For each hospital site: Baseline data will be collected for six months.
  **This extended beyond 6 months due to the COVID pandemic***
- Mobile Phone-administered Triage Tool (Experimental): For each hospital site: After the first six months of baseline data collection, the mobile phone-administered triage tool (or "Mobile Phone-based Triage Tool") will be implemented for a year.
  **This extended beyond 1 year due to the COVID pandemic***
  Interventions: Other: Mobile Phone-based Triage Tool

INTERVENTIONS:
Other: Mobile Phone-based Triage Tool — The proposed intervention is a mobile phone-administered survey. Participants that have been admitted to participating hospitals for treatment of injury will be contacted by mobile phone approximately two weeks after discharge. A seven-question survey will be administered over the phone to each participant. Cross-validation with a separately administered in-person physical exam will be performed to assess the survey tool's prediction of who needs further care for treatment of their injury.
  Arms: Mobile Phone-administered Triage Tool

SUMMARY:
After being admitted to and then discharged from a hospital in Cameroon for having experienced an injury, there is no established way for the health system to check in on how the discharged person is doing. The investigators have developed a set of questions with the hope that asking these questions--over the phone--to those who have been discharged from the hospital will allow them to determine which post-discharge patients would benefit from further care. The investigators believe that asking these questions over the phone is a good way of determining which post-discharge trauma patients would benefit from further care.

DETAILED DESCRIPTION:
Broadly, this study aims to answer three questions. (1) Is it feasible to call discharged trauma patients on their mobile phones to check up on them? (2) Can a defined set of questions help determine which discharged trauma patients require further medical care (and which discharged trauma patients do not require further medical care)? (3) Will checking in on discharged trauma patients reduce their experience of disability and economic consequences?

If an individual was a trauma patient who was admitted at and then discharged from one of the study's partner hospitals in Cameroon, the discharged individual (hereafter referred to as "the participant') will be receiving phone calls from one of the study's research assistants at the following post-discharge timepoints: 2 weeks, 1 month, 3 months, and 6 months. Whether the research assistant administers the defined set of questions developed by the study's investigators (see question 2, above) will depend on when the participant was discharged from the hospital. Regardless, all participants will be asked other important questions about the injury and any associated disabilities and economic consequences.

ELIGIBILITY:
Inclusion Criteria:

* All trauma registry patients at participating hospitals who provided cellphone numbers and are alive at hospital discharge are eligible for inclusion regardless of age, injury severity, or hospital disposition status.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3990 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Juillard, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (4):
- Cameroon (4):
  - Laquintinie Hospital, Douala
  - Edea Regional Hospital, Edéa
  - Limbé Regional Referral Hospital, Limbe
  - Pouma Catholic Hospital, Pouma

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome measures will be made available upon reasonable request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between August 5, 2019 and August 31, 2022. The baseline phase transitioned to intervention phase on Feb 16, 2020 at the 1st hospital with the planned step-wedge design. However, due to COVID restrictions in Cameroon to ensure participant safety, the study returned to baseline on April 27, 2020 and intervention phase restarted on Sep 7, 2020 while scrapping stepwedge design. Due to low recruitment numbers in COVID, study period was extended beyond the pre-specified 1 year.
Groups:
- No Mobile Phone-administered Triage Tool: For each hospital site: Baseline data will be collected for six months.
  **This extended beyond 1 year due to the COVID pandemic***
- Mobile Phone-administered Triage Tool: For each hospital site: After the first six months of baseline data collection, the mobile phone-administered triage tool (or "Mobile Phone-based Triage Tool") will be implemented for a year.
  **This extended beyond 1 year due to the COVID pandemic***
  Mobile Phone-based Triage Tool: The proposed intervention is a mobile phone-administered survey. Participants that have been admitted to participating hospitals for treatment of injury will be contacted by mobile phone approximately two weeks after discharge. A seven-question survey will be administered over the phone to each participant. Cross-validation with a separately administered in-person physical exam will be performed to assess the survey tool's prediction of who needs further care for treatment of their injury.
Period: Overall Study
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Started | 1491 | 2499
Completed | 837 | 1514
Not Completed | 654 | 985
Not completed — Death | 40 | 49
Not completed — Not reached on phone/ Did not consent | 614 | 936

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool | Total
Number analyzed (Participants) | 837 | 1514 | 2351
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Missing data: Information not provided, missing data not included in the analysis.
  years
    number analyzed (Participants) | 837 | 1513 | 2350
    (all) | 32 [24 to 43] | 32 [24 to 43] | 32 [24 to 43]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data: Information not provided, missing data not included in the analysis.
  Participants
    number analyzed (Participants) | 836 | 1512 | 2348
    Female | 246 | 351 | 597
    Male | 590 | 1161 | 1751
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants] — Population: Missing data: Information not provided, missing data not included in the analysis.
  Participants
    number analyzed (Participants) | 813 | 1511 | 2324
    No formal Education | 45 | 34 | 79
    Primary School | 199 | 308 | 507
    Secondary/High School | 431 | 866 | 1297
    Tertiary-University | 100 | 231 | 331
    Other | 38 | 72 | 110
Occupation [Count of Participants; unit: Participants] — Population: Missing data: Information not provided, missing data not included in the analysis.
  Participants
    number analyzed (Participants) | 833 | 1510 | 2343
    Housewife or husband | 66 | 80 | 146
    Salaried Worker | 199 | 310 | 509
    Self-Employed | 279 | 495 | 774
    Student | 115 | 189 | 304
    Unemployed (able to work) | 44 | 80 | 124
    Unemployed (unable to work) | 6 | 7 | 13
    Retired | 14 | 44 | 58
    Other | 110 | 305 | 415
Study site [Count of Participants; unit: Participants]
  Catholic Hospital Pouma | 85 | 122 | 207
  Laquintinie Hospital of Douala | 390 | 677 | 1067
  Edea Regional Hospital | 140 | 151 | 291
  Limbe Regional Hospital | 222 | 564 | 786
Injury location [Count of Participants; unit: Participants] — Population: Missing data: Information not provided, missing data not included in the analysis.
  Participants
    number analyzed (Participants) | 830 | 1507 | 2337
    Farm | 24 | 43 | 67
    Home | 90 | 151 | 241
    Road/Highway | 647 | 1203 | 1850
    Trade/Service Area | 17 | 20 | 37
    Industrial Construction | 18 | 35 | 53
    Other | 34 | 55 | 89
Injury mechanism [Count of Participants; unit: Participants] — Population: Missing data: Information not provided, missing data not included in the analysis.
  Participants
    number analyzed (Participants) | 832 | 1507 | 2339
    Road Traffic Injury | 601 | 1124 | 1725
    Stab/cut | 63 | 91 | 154
    Struck/hit by person | 49 | 81 | 130
    Fall | 73 | 140 | 213
    Other | 46 | 71 | 117

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Successful Contacts
Description: The number of successful contacts will be divided by the total number of contacts. A "successful" contact is when an enrolled patient answered the phone, and consented to the research assistant administering the questionnaire(s) planned for that phone call.
Time Frame: 2 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 1491 | 2499
Participants | 837 | 1514

2. Primary Outcome: Median Number of Attempts Required to Achieve a Successful Contact
Description: This is the median number of call attempts made until a research assistant is able to successfully administer the questionnaire(s) planned for that phone call.
Time Frame: 2 weeks after enrollment
Population: There was missing data for this variable hence the discrepancy between the overall number of participants analyzed for this variable and participants in the study. Missing data were dropped from the analysis.
Measure: Median (Inter-Quartile Range); unit: Number of calls
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 825 | 1476
Number of calls | 1 [1 to 1] | 1 [1 to 1]

3. Primary Outcome: Median Cost Associated With Personnel Time
Description: This measure is median monthly costs incurred to pay the research assistant for the time s/he spends making the required phone calls per patient.
Time Frame: At the end of the study (2 weeks after the 2-year intervention phase (extended due to COVID))
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 1491 | 2499
Dollars | 3.75 [2.21 to 4.87] | 3.56 [3.04 to 5.18]

4. Primary Outcome: Median Cost Associated With Telephone Time
Description: This measure is the median costs incurred to make phone calls per patient in each study phase.
Time Frame: At the end of the study (2 weeks after the 2-year intervention phase (extended due to COVID))
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 1491 | 2499
Dollars | 2.89 [2.42 to 4.43] | 4.92 [4.24 to 5.67]

5. Primary Outcome: Telephone Triage Tool Administration Time
Description: This measure will be calculated based on how much time it takes to administer the telephone triage tool.
Time Frame: After administration of the telephone triage tool (i.e. about 2 weeks after enrollment)
Population: Telephone triage tool was the "intervention" and was only administered in the intervention phase. There was missing data for this variable hence the discrepancy between the overall number of participants analyzed for this variable and participants in the study. Missing data were dropped from the analysis.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 0 | 1510
seconds |  | 81.5 [48 to 146]

6. Primary Outcome: Physician Assessment of Whether a Patient Would Benefit From Further Services
Description: This is a binary measure. After a physician examines a participant, s/he will determine whether s/he thinks the participant would benefit from further services (including additional follow-up care, and/or diagnostic or therapeutic interventions).
Time Frame: Immediately after the physician administers the physical exam (i.e. about 3 weeks after enrollment)
Population: Physician examination occurred only in the intervention phase where participants who were administered the telephone triage tool were asked to return for a physician examination to cross-validate tool finding. The number analyzed represents the number of patients who returned for the physician examination.
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 0 | 560
Participants
  Yes |  | 323
  No |  | 237

7. Primary Outcome: Physician Assessment of Whether a Patient Was at Moderate to High Risk for a Poor Outcome (HR) Without Additional Intervention
Description: After a physician examines a participant, s/he will determine whether s/he thinks the participant is at low, moderate or high risk for a poor outcome (HR) without additional intervention using subjective clinical assessment.
Time Frame: Immediately after the physician administers the physical exam (i.e. about 3 weeks after enrollment)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 0 | 560
Participants
  Low risk |  | 357
  Moderate risk |  | 160
  High risk |  | 43

8. Primary Outcome: Triage Risk Score (TRS)
Description: To develop a sensitive model capable of risk stratifying triaged patients for high risk (HR), all candidate questions from the telephone triage tool found to associate with HR on univariate regression were weighted by their predictive coefficient and added to generate a triage risk score (TRS) ranging from a minimum score of 0 (lowest risk) to a maximum possible score of 43.9 (highest risk). Triage Risk Score (TRS) less than or equal to 1.3 (1st quartile) was designated as low risk, TRS 1.4 to 4.0 (2nd & 3rd quartile) as moderate risk, and TRS greater than or equal to 4.1 (fourth quartile) as high risk.
Time Frame: At the end of intervention phase (about 1 year after enrollment).
Population: The telephone triage tool was administered only in the intervention phase. The number analyzed represents the subset of patients who returned for the physician examination.
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 0 | 560
Participants
  Low risk |  | 220
  Moderate risk |  | 217
  High risk |  | 123

9. Primary Outcome: Acceptability Score of Mobile Phones as a Follow-up Tool
Description: This is a numerical measure that represents the sum of the positive responses that participants give to each question that assesses the acceptability of mobile phones as a follow-up tool. The scale for the acceptability score of mobile phones as a follow-up tool ranges from 0 to 6, where 0 means the participant's responses indicate the participant believes mobile phones are definitely not an acceptable follow-up tool and 6 means the participant's responses indicate the participant believes mobile phones are definitely an acceptable follow-up tool.
Time Frame: 2 weeks after enrollment
Population: The acceptability tool was administered to a subset of patients.
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 218 | 962
Participants
  Score of 1 | 1 | 0
  Score of 2 | 0 | 3
  Score of 3 | 3 | 11
  Score of 4 | 10 | 28
  Score of 5 | 30 | 175
  Score of 6 | 174 | 745

10. Primary Outcome: Proportion of Injured Patients Who Seek Clinical Follow-up Evaluation
Description: This will be calculated as follows: The denominator will be the number of discharged trauma patients enrolled in the study. The numerator will be the number of discharged trauma patients enrolled in the study who seek any clinical follow-up evaluation at the 2 weeks post-discharge phonecall.
Time Frame: After the 2week post-discharge phonecall.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 776 | 946
Participants | 409 | 615

11. Secondary Outcome: Glasgow Outcomes Scale-Extended (GOSE) Disability Level
Description: The GOSE disability level that participants in the study report. For each participant, GOSE disability level will be determined using the augmented GOSE (aGOSE) instrument, which assesses factors like the participant's independence inside and outside the home, work, social and leisure activities, family and friendship, etc. Each time after administration of the aGOSE instrument, the participant's GOSE disability level will be calculated. The aGOSE score is reported for the 2-week post-discharge timepoint.
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories (worse to best respectively): Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery. The Extended GOS (GOSE) which was used in this study provides more detailed categorization into eight categories by subdividing the categories of severe disability, moderate disability and good recovery into a lower and upper category.
Time Frame: At the 2week post-discharge telephone phonecall.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 831 | 968
Participants
  Upper good recovery | 175 | 148
  Lower good recovery | 77 | 163
  Upper moderate disability | 42 | 77
  Lower moderate disability | 76 | 52
  Upper severe disability | 227 | 349
  Lower severe disability | 179 | 160
  Vegetative State | 15 | 0
  Death | 40 | 19

12. Secondary Outcome: Economic Consequences of Injury: Did it Become More Difficult for the Family to Afford Expenses Such as Food and Rent?
Description: Participants were asked if following the injury it became more difficult for the family to afford expenses such as food and rent.
Time Frame: At the 2week post-discharge telephone phonecall.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 724 | 918
Participants
  Yes | 524 | 768
  No | 200 | 150

13. Secondary Outcome: Economic Consequences of Injury: Did the Family Spend Saved Money?
Description: Participants were asked if following the injury the family had to spend their savings.
Time Frame: At the 2week post-discharge telephone phonecall.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 837 | 989
Participants
  Yes | 601 | 890
  No | 236 | 99

14. Secondary Outcome: Economic Consequences of Injury: Did the Family Borrow Money?
Description: Participants were asked if following the injury the family had to borrow money to meet up with expenses.
Time Frame: At the 2week post-discharge telephone phonecall.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
Number analyzed (Participants) | 837 | 989
Participants
  Yes | 370 | 476
  No | 467 | 513

ADVERSE EVENTS:
Time Frame: At the 2 weeks post-discharge phone call.
Description: During an answered post-discharge phone call, respondents were asked on the survey if injured patient was alive.
Arm/Group | No Mobile Phone-administered Triage Tool | Mobile Phone-administered Triage Tool
All-Cause Mortality (participants affected / at risk) | 40/1491 | 49/2499
Serious Adverse Events (participants affected / at risk) | 0/1491 | 0/2499
Other Adverse Events (participants affected / at risk) | 0/1491 | 0/2499

LIMITATIONS AND CAVEATS:
Early in the COVID pandemic due to restrictions in Cameroon and to ensure safety of participants, changes were made such as pausing intervention phase where patients were asked to return to the hospital for a physician exam to cross-validate the telephone triage tool and reverting to baseline. The step-wedge design was also scrapped as this was disrupted by the pause. Low recruitment numbers in COVID also accounted for the intervention phase to be extended beyond the pre-specified timeline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03805646/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT03805646/ICF_001.pdf